CLINICAL TRIAL: NCT06751134
Title: A Study to Evaluate the Safety, Preliminary Efficacy, Pharmacokinetics of CNK-UT Cells to Treat the Patients with Relapsed/refractory Neuroblastoma
Brief Title: Chimeric Natural Killer Receptor-Universal T Cells for Relapsed or Refractory Neuroblastoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing Children's Hospital (Other)
Responsible Party: Principal Investigator, Fang Yongjun, Prof., Nanjing Medical University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNK-UT-IIT202304
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Neuroblastoma, Recurrent, Refractory
Keywords: Chimeric natural killer receptor universal T-cells, relapsed/refractory Neuroblastoma
MeSH Terms: conditions — Neuroblastoma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CNK-UT cells therapy (Experimental): 1. Dose Escalation： Single-dose intravenous injection of CNK-UT cells (3~34×10^7 CNK+ cells/kg).
  2. Dose Expansion:
  Multiple-dose intravenous injection of CNK-UT cells according to the results of dose escalation.
  Interventions: Drug: Chimeric Natural Killer Receptor Universal T-cells (CNK-UT)

INTERVENTIONS:
Drug: Chimeric Natural Killer Receptor Universal T-cells (CNK-UT) — OUTLINE: This is a dose-escalation study of CNK-UT cells followed by a dose-expansion study.
  1. Dose Escalation (Single Ascending Dose Study, SAD): During SAD study stage, the participants will be intravenous infused with CNK-UT cells (3~34×10^7 CNK+ cells/kg)with a"3 +3" design to determine the maximum tolerated dose. During single ascending dose (SAD) study stage, the participants will receive a single dose of CNK-UT cells before the DLT observation period (21 days). If the participants do not experience DLT, they will be able to enter a multiple ascending dose (MAD) study stage.
  2. Dose Expansion (multiple ascending dose study, MAD): During MAD study stage, the participants will receive multiple doses of CNK-UT cells. The dosage and frequency of drug administration in the dose expansion stage can be adjusted and determined according to the SAD study.

SUMMARY:
This is a single arm, open-label, multi-center, pilot studies (Investigator Initiated Trial, IIT) to evaluate the safety, preliminary efficacy, pharmacokinetics of universal T-cells engineered with chimeric natural killer receptor (CNK-UT) to treat the patients with relapsed/refractory Neuroblastoma.

DETAILED DESCRIPTION:
This is a single arm, open-label, phase I, dose escalation/dose expansion study to assess the safety of CNK-UT cells therapy, and to obtain the preliminary efficacy and pharmacokinetics result in participants who have been diagnosed with relapsed/refractory Neuroblastoma.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 1-12 years with weight≥10kg, male or female;
2. The child and/or guardian has signed the informed consent form (ICF) and has the ability to comply with the study requirements.
3. Diagnosed with relapsed/refractory neuroblastoma. Clinical diagnostic criteria and first-line standard treatment can refer to the NCCN guidelines:

   1. Relapsed neuroblastoma: New lesions appear at the primary site or other locations 4 weeks after achieving complete remission through first-line standard treatment.
   2. Refractory neuroblastoma: Failure to achieve complete remission after standard treatment protocols, which include induction chemotherapy, surgery, and radiotherapy targeting the primary tumor and residual metastatic sites;
4. Prior to enrollment, appropriate measures can be implemented to ensure that the subject's disease status is either partial remission (PR) or stable disease (SD).
5. According to the INRC efficacy criteria, there must be at least one lesion whose efficacy can be assessed through functional imaging (123I-MIBG) and/or bone marrow examination (bone marrow aspiration or biopsy). If soft tissue lesions are present, the longest diameter of the target lesion should be ≤2 cm.
6. Tumor tissue sections or paraffin blocks can be provided, and it has been confirmed through immunohistochemistry (IHC) that the tumor tissue expresses B7-H3.
7. Lansky score>60；
8. Estimated life expectancy > 12 weeks;
9. Adequate organ and bone marrow function, and the laboratory test value meets the following requirements within 7 days before enrollment, as follows:

(1)Blood Routine Test: Absolute neutrophil count(ANC)≥1.5×10^9/L;Absolute lymphocyte count (ALC)≥0.2×10^9/L；Platelet count ≥75×10^9/L; Haemoglobin≥90g/L; (2)Heart: Left ventricular ejection fraction (LVEF)≥50%;Cardiac function Grade I-II; (3)Pulmonary function: indoor oxygen saturation≥92%. (4)Hepatic function：Total bilirubin≤3×ULN; Aspartate aminotransferase (AST) or alanine aminotransferase (ALT)≤5×ULN; (5)Renal function: Serum creatinine≤2×ULN, or Creatinine clearance rate (CCR)≥60 mL/min (Cockroft-Gault formula); 10.All toxic responses originating from previous radiotherapy, chemotherapy, or other treatments (occurring within 4 weeks or 5 half-lives of anti-tumor drugs therapy [including but not limited to chemotherapy, targeted therapy, immunotherapy, Chinese herbal medicine]) have returned to NCI CTCAEV5.0 Grade≤1 (except for hair loss).

Exclusion Criteria:

1. Suffering from malignant tumors or diagnosed within 5 years before enrollment, excluding radical skin basal cell carcinoma, skin squamous cell carcinoma, thyroid cancer, breast cancer (ductal carcinoma in situ) and / or radical resection of carcinoma in situ.
2. Participants with symptomatic central nervous system (CNS) metastasis confirmed by imaging or pathological examination.
3. Participants with MIBG non-avid disease.
4. Participants with a history of organ transplantation（excluding stem cell transplantation）;
5. Participants with active autoimmune diseases requiring systemic treatment (such as the use of disease-modifying drugs, corticosteroids, or immunosuppressants) are considered. The use of replacement therapies (such as thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency) is permitted. A known history of primary immunodeficiency is also noted. For patients who only test positive for autoimmune antibodies, the presence of autoimmune disease must be confirmed based on the investigator's judgment.
6. Uncontrolled or irreparable systemic diseases, metabolic disorders, or other non-malignant organ diseases or cancer sequelae, which may lead to higher medical risks and/or uncertainties in survival assessment.
7. Active pulmonary tuberculosis (TB), who is receiving anti-tuberculosis treatment or has received anti-tuberculosis treatment within 1 year before enrollment; human immunodeficiency virus (HIV) infection, known syphilis infection.
8. Severe infections that are either active or poorly controlled clinically within 4 weeks prior to enrollment, including but not limited to hospitalization due to infections, bacteremia, or severe pneumonia complications (excluding mild urinary tract infections and upper respiratory tract infections).
9. Received radiotherapy, chemotherapy (excluding lymphodepletion), molecular targeted therapy, immune checkpoint inhibitors, or other anti-tumor treatments within 4 weeks or 5 half-lives (whichever is shorter) before cell infusion..
10. Participants who have undergone major surgery (craniotomy, thoracotomy, or laparotomy) within 4 weeks prior to the initiation of the study, or have severe unhealed wounds, ulcers, or fractures.
11. Participants who have received treatment from other clinical trials within 4 weeks prior to the initiation of the study.
12. Participants who receive attenuated live vaccines within 4 weeks prior to the initiation of the study.
13. Participants who have used any gene therapy products prior to cell infusion.
14. Allergic to components of CNK-UT injection.
15. Participants suffer from known mental or substance abuse disorders, which may interfere with their ability to comply with research requirements.
16. Participants considered by the investigator to have other potentially life-threatening serious complications that may interfere with the evaluation of this study..
17. Other situations that the participant is identified by the investigator as unsuitable to participate in the study.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2024-12-28 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Related adverse events (AEs) | up to 1 year
  Incidence of Treatment Related AEs, AEs of special interest and serious adverse events (SAEs) assessed by NCI-CTCAE v5.0 criteria

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 1 year
  Overall response is defined as either a complete or partial response (CR+PR), the response should be confirmed no less than 4 weeks after the first evaluation.
Duration of Response (DOR) | up to 1 year
  The period from the first evaluation of CR or PR to the first evaluation of PD or death of any cause.
Disease control rate (DCR) | up to 1 year
  The number of cases in which response are achieved from the start of cells infusion/the total number of evaluable cases (%).
Progression-free Survival (PFS) | up to 1 year
  The period from the day when the participant receives the cell therapy to the first recorded disease progression (whether treated or not) or death of any cause, which occurs first.
Overall survival (OS) | up to 1 year
  The period from the first infusion to any cause of death.
Pharmacokinetics (PK) (Cmax) | up to 1 year
  The Peak Plasma concentration (Cmax) of amplified CNK-UT DNA in peripheral blood after infusion.
Pharmacokinetics (PK) (Tmax) | up to 1 year
  The time to reach the maximum concentration (Tmax).

OTHER OUTCOMES:
biomarkers | up to 1 year
  Ferritin, lactate dehydrogenase (LDH), neuron specific enolase (NSE) will be analyzed.
Levels of peripheral blood lymphocyte subsets | up to 1 year
  Percentage of T cell、B cell、NK Cells、Treg cell and MDSC in peripheral blood detected by FCM after infusion.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Nanjing Children's Hospital, Nanjing, Jiangsu
  - Nanjing, Nanjing, Jiangsu